CLINICAL TRIAL: NCT00516516
Title: Oral L-Carnitine for the Treatment of Muscle Cramps in Pregnancy: A Randomized, Controlled Trial
Brief Title: Oral Carnitine for Cramps in Pregnancy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low interest in study, slow recruitment
Sponsor: University of Southern California (Other)
Collaborators: Health Research Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-06-00233
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2009-10

CONDITIONS: Muscle Cramp
Keywords: muscle cramp; pregnancy; carnitine; randomized controlled clinical trials
MeSH Terms: conditions — Muscle Cramp | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I (Experimental): Oral L-Carnitine, 1g PO twice daily
  Interventions: Dietary Supplement: L-Carnitine
- II (Placebo Comparator): Placebo, similar in appearance to experimental drug, given orally twice daily.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-Carnitine — L-Carnitine, 1g orally, twice daily
  Arms: I
Dietary Supplement: Placebo — Placebo, similar in appearance to study tablets, given orally, twice daily.
  Arms: II

SUMMARY:
Muscle cramps occur frequently among pregnant women, and few therapeutic options exist. This is a study of oral L-carnitine, a dietary supplement, for the treatment of muscle cramps in pregnancy. Our hypothesis is that carnitine will alleviate or eliminate muscle cramps experienced by pregnant women.

DETAILED DESCRIPTION:
Muscle cramps occur frequently among pregnant women, and few therapeutic options exist. This is a study of oral L-carnitine, a dietary supplement, for the treatment of muscle cramps in pregnancy. The conceptual basis for this study comes from the fact that carnitine has been used effectively in multiple randomized trials for the treatment of muscle cramps in other carnitine deficient states (such as hemodialysis). In pregnancy, women have decreased serum carnitine concentrations (from decreased intake, increased clearance by the kidney, and increased demands from the fetus). Thus, our hypothesis is that carnitine will alleviate or eliminate muscle cramps experienced by pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 or older
* Gestational Age 12 to 33 weeks
* Occurrence of muscle cramps at least once weekly
* Ability to tolerate oral L-Carnitine
* Ability / willingness to provide informed consent in English or Spanish

Exclusion Criteria:

* Prior treatment for muscle cramps during this pregnancy
* Chronic muscle cramps prior to pregnancy
* Magnesium administration beyond that contained in prenatal vitamins
* History of seizures
* History of Pre-term delivery before 36 weeks gestational age
* Inability to tolerate oral L-Carnitine (e.g. hyperemesis gravidarum)
* Inability or unwillingness to provide informed consent

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-07; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Complete elimination of muscle cramps | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Emiliano R Chavira, MD,MPH, Principal Investigator — University of Southern California, Keck School of Medicine, Division of Maternal-Fetal Medicine; Thomas M Goodwin, MD, Principal Investigator — University of Southern California, Keck School of Medicine, Division of Maternal-Fetal Medicine
Locations (2):
- United States (2):
  - USC Perinatal Group Medical Office, Los Angeles, California
  - Women's & Children's Hospital Midwife Clinic, Los Angeles, California